CLINICAL TRIAL: NCT05112185
Title: Healthy Drinks, Healthy Futures: The Impact of a Childcare-based Healthy Beverages Intervention on Young Children's Food and Beverage Intake and Obesity
Brief Title: Childcare Healthy Beverage Access, Food and Beverage Intake, and Obesity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, San Francisco (Other); University of California Agriculture and Natural Resources (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Anisha I Patel, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 61606; 1R01DK127124-01A1 (NIH)
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: water; sugar-sweetened beverages; childcare
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Beverage Access and Promotion (Experimental): Intervention group will receive BPA-free self-serve pitchers and cups for serving water at mealtimes, individualized education to help families set healthy drinks goals for their family, and a curricula focused on increasing intake of water and healthy beverages.
  Interventions: Behavioral: Healthy Drinks, Healthy Futures
- Control (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Healthy Drinks, Healthy Futures — The Healthy Drinks, Healthy Futures intervention consists of increased access to healthy beverages in childcare centers and education directed to children and their families to increase the intake of healthy beverages, including motivational beverage counseling for families and lessons for children in childcare centers.
  Arms: Healthy Beverage Access and Promotion

SUMMARY:
Interventions that promote water consumption in place of sugar-sweetened beverages have shown promise for preventing childhood obesity in schoolchildren. Yet to date, no studies have examined whether applying this approach in childcare centers could help to prevent childhood obesity at an even earlier stage of development. This cluster-randomized controlled trial will fill gaps by examining how a multilevel childcare-based healthy beverage intervention affects young children's consumption of beverages and obesity.

DETAILED DESCRIPTION:
There is little debate that sugar-sweetened beverages (SSBs; drinks with added sugar) lack nutrition, are a major source of added sugar and calories, and promote obesity and poor cardiometabolic health, especially when consumed during early childhood. Nearly half of children aged 2-5 drink SSBs on a daily basis, with heavier consumption in low-income Latino children. After decades of research, it is clear that there is no single "magic bullet" for solving obesity. What we need are bundled interventions that combine incremental changes that transform food environments with targeted behavior changes that steer people towards those healthy options. Childcare centers, which serve 12.5 million children per year, provide an efficient way to intervene early by engaging childcare providers and parents to make resonant, mutually reinforcing changes in both the home and childcare environment. Interventions that promote water consumption in place of SSBs have shown promise for preventing childhood obesity in schoolchildren. Yet, no studies have examined whether interventions to promote intake of water instead of SSBs in childcare could prevent childhood obesity at an even earlier stage of development. The proposed cluster-randomized controlled trial will test the efficacy of an intervention called Healthy Drinks, Healthy Futures (Bebidas Saludables, Futuros Saludables) that is culturally adapted for Latino children and families. Following the Social-Ecological Model and Social Learning Theory, the intervention supports complementary changes in the childcare and home food environments that promote water consumption while reducing SSB availability. This is combined with education for childcare providers and children, and a one-on-one brief motivational counseling intervention with parents to reduce SSB intake and encourage water consumption in the home. Fourteen childcare centers serving low-income, predominately Latino children (n=420) will participate in this trial. The primary outcome is child BMI z-score (BMI standard deviation score). Key secondary outcomes are intake of water and beverage calories at centers and at home. Outcomes will be captured using anthropometrics (weight, height), and beverage frequency questionnaires at baseline, 6-months, and 12-months post-intervention. Plate waste measurements (water and caloric intake at centers) and Automated Self-Administered 24-hour dietary recalls (water and caloric intake at home) will occur at baseline and 12 months post-intervention. Surveys of childcare providers and parents will allow us to explore possible mediators of the intervention effect. We hypothesize that the childcare-based healthy beverage intervention will increase intake of water and reduce beverage calories consumed at both childcare and at home. BMI z-score will also improve among children in intervention centers vs. control centers. If shown to be effective, the Healthy Drinks, Healthy Futures intervention will offer a strategy for intervening early to prevent obesity for millions of low-income children attending childcare centers. Findings from this study will contribute to the science of multilevel obesity prevention, and inform the implementation of state, federal, and local policies to promote healthy beverage intake in childcare centers.

ELIGIBILITY:
Inclusion Criteria:

* Preschool-age children and families who don't have health conditions that preclude intake of water

Exclusion Criteria:

* Children not of preschool-age
* Children and families who do not speak English or Spanish

Ages: 2 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 882 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in BMI z-score | Baseline, 6-months, and 12-months after the start of the study.
  The BMI measure will be calculated using height and weight measurements.

SECONDARY OUTCOMES:
Total caloric intake from beverages at childcare centers | Baseline and 12-months after the start of the study.
  Plate waste measurements will be used to calculate total daily caloric intake from beverages at childcare centers.
Total beverage caloric intake from beverages at home | Baseline and 12-months after the start of the study.
  Automated Self-Administered 24-Hour (ASA24) will be used to calculate total daily caloric intake from beverages at home.
Beverage intake frequency | Baseline, 6-months, and 12-months after the start of the study.
  BevQ 19 and BevQ PS

CONTACTS AND LOCATIONS:
Overall Officials: Anisha Patel, MD, MSPH, Principal Investigator — Stanford University
Locations (1):
- Stanford, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No